CLINICAL TRIAL: NCT00000155
Title: The Collaborative Longitudinal Evaluation of Keratoconus (CLEK) Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Eye Institute (NEI) (NIH)
Other Study IDs: NEI-57
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-11

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
To describe the clinical course of keratoconus and to describe the relationships among its visual and physiological manifestations, including high- and low-contrast visual acuity, corneal curvature, slit lamp biomicroscopic findings, corneal scarring, and quality of life.

To identify risk factors and protective factors that influence the severity and progression of keratoconus.

DETAILED DESCRIPTION:
Keratoconus is a bilateral, asymmetric, chronic, progressive ectasia of the cornea characterized by steepening and distortion of the cornea, thinning of the apical cornea, corneal scarring, and treatment-related sequelae, such as abrasions from contact lenses and surgical complications. Patients experience distorted vision that worsens with disease progression. Their vision is typically corrected with spectacles early in the disease and, later, with rigid contact lenses. Some patients eventually undergo corneal transplantation in one or both eyes. Keratoconus affects people in their prime earning years and profoundly affects their lives.

Previous large-scale studies of keratoconus have focused on incidence and prevalence, etiologies, or the clinical management of keratoconus. Few have characterized the course of the disease and risk factors for its progression in large samples of keratoconus patients. The incidence of vision-threatening corneal scarring in keratoconus is unknown. Patient's most frequent questions--how rapidly their keratoconus will progress, how bad their vision will become, whether they will need corneal surgery, how successful their contact lenses will be--cannot be answered on the basis of the current body of knowledge.

The need for a prospective, observational study of keratoconus patients is great. Results from this study will address keratoconus patient's unanswered questions and will enable eye care practitioners to manage this complex ocular disease better.

The Collaborative Longitudinal Evaluation of Keratoconus (CLEK) Study is a multicenter, observational study of 1,209 keratoconus patients followed for 3 years.

Patients are examined annually. Study measures include visual acuity, patient-reported quality of life, manifest refraction, keratometry, photodocumentation of the cornea to identify central corneal scarring, photodocumentation of the flattest contact lens that just clears the cornea, slit lamp biomicroscopy, and corneal topography. In rigid contact lens wearers, the fluorescein pattern of the patient's habitual contact lenses is photodocumented.

Patients are examined at 15 clinical centers. The clinical centers enrolled 1,209 patients in 12 months.

ELIGIBILITY:
Patients with keratoconus were eligible if they were at least 12 years old; had an irregular cornea as determined by keratometry, retinoscopy, or direct ophthalmoscopy in at least one eye; had Vogt's striae, Fleischer's ring, or corneal scarring characteristic of keratoconus in at least one eye; and planned to stay in the area for at least 3 years. They were ineligible if they had bilateral corneal transplants or bilateral nonkeratoconic eye disease (cataract, intraocular lenses, macular disease, or optic nerve disease other than glaucoma).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-06

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - University of California, Berkeley, School of Optometry, Berkeley, California
  - Southern California College of Optometry, Fullerton, California
  - Jules Stein Eye Institute, University of California at Los Angeles, Los Angeles, California
  - Nova Southeastern University, Health Professions Division, College of Optometry, Fort Lauderdale, Florida
  - University of Illinois at Chicago, Department of Ophthalmology and Visual Sciences, Chicago, Illinois
  - Indiana University, School of Optometry, Bloomington, Indiana
  - University of Missouri-St. Louis, School of Optometry, St Louis, Missouri
  - SUNY State College of Optometry, New York, New York
  - University Hospitals of Cleveland, Department of Ophthalmology, Cleveland, Ohio
  - The Ohio State University, College of Optometry, Columbus, Ohio
  - Pennsylvania College of Optometry, The Eye Institute, Philadelphia, Pennsylvania
  - Northeastern Eye Institute, Scranton, Pennsylvania
  - University of Utah, John Moran Eye Center, Salt Lake City, Utah
  - Gundersen Lutheran, La Crosse, Wisconsin

REFERENCES:
- [Background] Barr JT, Gordon MO, Zadnik K, Pellican K, Edrington TB. Photodocumentation of corneal scarring. Collaborative Longitudinal Evaluation of Keratoconus Study Group. J Refract Surg. 1996 May-Jun;12(4):492-500. doi: 10.3928/1081-597X-19960501-13. PMID 8771545
- [Background] Edrington TB, Barr JT, Zadnik K, Davis LJ, Gundel RE, Libassi DP, McMahon TT, Gordon MO. Standardized rigid contact lens fitting protocol for keratoconus. Optom Vis Sci. 1996 Jun;73(6):369-75. doi: 10.1097/00006324-199606000-00003. PMID 8807647
- [Background] Gundel RE, Libassi DP, Zadnik K, Barr JT, Davis L, McMahon TT, Edrington TB, Gordon MO. Feasibility of fitting contact lenses with apical clearance in keratoconus. Optom Vis Sci. 1996 Dec;73(12):729-32. doi: 10.1097/00006324-199612000-00002. PMID 9002088
- [Background] Zadnik K, Barr JT, Gordon MO, Edrington TB. Biomicroscopic signs and disease severity in keratoconus. Collaborative Longitudinal Evaluation of Keratoconus (CLEK) Study Group. Cornea. 1996 Mar;15(2):139-46. doi: 10.1097/00003226-199603000-00006. PMID 8925661